CLINICAL TRIAL: NCT02476201
Title: Quartet Lead and Resynchronization Therapy Options - Assessing the Response Rate at 6 Months in CRT Patients Implanted With a Quartet Left Ventricular(LV) Quadripolar Lead and the MultiPoint Pacing (MPP) Feature Activated
Brief Title: Quartet Lead and Resynchronization Therapy Options III (QUARTO_III)
Acronym: QUARTO_III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD_789
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac Resynchronization Therapy; Quadripolar Left Ventricular Lead; Multipoint Pacing; Hemodynamic Response
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MPP ON (Experimental): To activate the Multipoint Pacing (MPP) feature to ON in all patients
  Interventions: Device: MPP ON

INTERVENTIONS:
Device: MPP ON — Patients implanted with a Cardiac Resynchronization Therapy CRT-D device and a Quartet Left Ventricular (LV) quadripolar lead and with the MultiPoint Pacing (MPP) feature activated

SUMMARY:
The purpose of the study is to assess prospectively at 6 months the percentage of responder patients implanted with a Cardiac Resynchronization Therapy (CRT-D) device and a Quartet Left Ventricular (LV) quadripolar lead and with the MultiPoint Pacing (MPP) feature activated.

DETAILED DESCRIPTION:
The primary endpoint of the study is to measure prospectively at 6 months the percentage of responder* patients implanted with a Quartet LV quadripolar lead and with the MultiPoint Pacing feature activated compared with No Pacing at baseline.

*A positive CRT response is defined as an improvement of more than 15 % in Left Ventricular End Systolic Volume (LVESV) at 6 months post-implant, measured by Echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Patient that will be implanted with a Cardiac Resynchronization Therapy (CRT-D) with the MultiPoint Pacing (MPP) feature under the current Guidelines indications for CRT-D implant (including upgrades from single or dual chamber Defibrillator or Pacemaker).
* Patient that will be implanted with a Quartet Left Ventricular (LV) quadripolar lead.
* In sinus rhythm at baseline visit.
* Patients with Left Bundle Branch Block (LBBB)
* Must be willing and able to comply with study requirements.
* Older than 18 years
* Must indicate their understanding of the study and willingness to participate by signing an appropriate informed consent form.

Exclusion Criteria:

* Already has a CRT device implanted.
* Myocardial Infarction or unstable angina within 40 days prior the enrollment.
* New York Heart Association (NYHA) Class IV
* Recent cardiac revascularization in the 4 weeks prior to enrollment.
* Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) in the 3 months prior the enrollment.
* Classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 12 months.
* Primary valvular disease requiring surgical intervention.
* Atrial Fibrillation (AF):

  * Persistent AF at the time of enrollment or 30 days prior the enrollment
  * Permanent AF not treated with Atrio-Ventricular node ablation within 2 weeks after the CRT-D implant
  * History or incidence of Paroxysmal or Persistent AF within 30 days prior the enrollment
* Patient for whom suitable Transthoracic echocardiographic images for determining the cardiac output (CO) and LV volumes cannot be obtained.
* Undergone a cardiac transplantation or being waiting for it
* Life expectancy < 6 months
* Pregnancy or planning to become pregnant
* Unable to comply with the follow up schedule
* Currently participating in any other clinical investigation.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Sanz, Study Director — Abbott Medical
Locations (1):
- Hospital Virgen de la Victoria, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment began on 11-Feb-2016 and the last enrollment occurred on 13-Aug-2018.
Groups:
- MPP ON: Patients implanted with a Cardiac Resynchronization Therapy CRT-D device and a Quartet Left Ventricular (LV) quadripolar lead will be programmed with the MultiPoint Pacing (MPP) feature activated.
Period: Overall Study
Arm/Group | MPP ON
Started | 105
Implant Attempts | 103
Sucessful Implants | 102
6 Months Visit | 82
Completed | 79
Not Completed | 26
Not completed — Unable to program MPP | 9
Not completed — Study echo not performed | 5
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Lost to Follow-up | 2
Not completed — MPP programmed to OFF | 2
Not completed — Withdrawal by Subject | 1
Not completed — Unsuccessful implant | 1

BASELINE CHARACTERISTICS:
Groups:
- MPP ON: MPP ON: Subjects implanted with a Cardiac Resynchronization Therapy CRT-D device and a Quartet Left Ventricular (LV) quadripolar lead and with the MultiPoint Pacing (MPP) feature activated.
Arm/Group | MPP ON
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 97
  Portugal | 8
Left Ventricular End Systolic Volume (LVESV) [Mean (Standard Deviation); unit: mililiters] — Population: The number of subjects in this analysis population differs from the overall study population because LVESV was only calculated in the 77 analyzable subjects with 6-month echocardiogram data available.
  mililiters
    number analyzed (Participants) | 77
    (all) | 127.78 (48.87)
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — The NYHA provides a simple way of classifying the extent of heart failure:
  NYHA I: No limitation of physical activity. Ordinary physical activity does not cause fatigue, palpitation, dyspnea.
  NYHA II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  NYHA III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  NYHA IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest.
  Participants
    NYHA I | 6
    NYHA II | 60
    NYHA III | 39
    NYHA IV | 0
Cardiomyopathy Etiology [Count of Participants; unit: Participants]
  Non-ischemic | 61
  Ischemic | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of CRT Responders
Description: The number of CRT responders was evaluated at 6 months post-implant. A CRT responder patient was a patient with an improvement of >15 % in LVESV, as measured by echocardiography.
Time Frame: 6 months
Population: The analysis population included subjects implanted with a Quartet LV quadripolar lead and with the MPP feature activated and who had a 6-month CRT response evaluation via echocardiography. Subjects who withdrew prior to the 6-month visit, did not complete the 6-month visit, or had relevant 6-month data missing were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MPP ON
Number analyzed (Participants) | 79
Participants | 53
Statistical Analysis 1: Comparison: MPP ON; Test type: Superiority — Using a one-sided, one sample Exact Binomial Test and a significance level of 2.5%, the study required 74 patients to reach a power of 90%. With the MPP feature activated at baseline, it was assumed that the proportion of responders at 6 months was 75%. The MPP responder rate was compared to 57%, which is the responder rate obtained from literature for patients without the MPP feature activated; p = 0.0435, Exact binomial; Percentage = 67.1, 97.5% CI 1-sided [lower limit 55.6]

2. Secondary Outcome: Changes in LV Echocardiographic Parameters
Description: An echocardiogram was performed at baseline and at 6 months in subjects with MPP activated. The outcome evaluated the percentage of change in LVESV, left ventricular end-diastolic volume (LVEDV), left ventricular end systolic diameter (LVESD), left ventricular end diastolic diameter (LVEDD), and left ventricular ejection fraction (LVEF) as compared to baseline prior to implant.
  The values of change with positive numbers represent increases and negative numbers represent decreases.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MPP ON
Number analyzed (Participants) | 74
Percent change
  LVESV | -25.33 (31.42)
  LVEDV | -14.90 (28.09)
  LVESD | -10.72 (14.53)
  LVEDD | -7.23 (11.72)
  LVEF | 9.37 (12.2)

3. Secondary Outcome: Number of CRT Super-responders
Description: The outcome evaluated the number of CRT super-responders at 6 months in subjects with MPP activated. A super-responder is defined as a subject with a mean absolute LVEF increase of >14% at 6 months post-implant compared to baseline.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MPP ON
Number analyzed (Participants) | 77
Participants | 27

4. Secondary Outcome: Rates of Hospitalization and Mortality
Description: The outcome measures rates of all-cause mortality, all-cause hospitalization, cardiovascular hospitalization, and heart failure hospitalization. In addition, the outcome measures the combined endpoint of mortality and heart failure hospitalization and mortality and cardiovascular hospitalization. For the combined endpoints, if a participant experienced both endpoints, they were counted as one participant.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- All Enrolled Subjects: All subjects enrolled in the study are included in this outcome measure.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 105
Participants
  All-cause mortality | 2
  All-cause hospitalization | 12
  Heart failure hospitalization | 1
  Cardiovascular hospitalization | 4
  Combined mortality/heart failure hospitalization | 2
  Combined mortality/cardiovascular hospitalization | 6

5. Secondary Outcome: Change in NYHA Classification
Description: The outcome measures status changes in NYHA classification at 6 months for subjects with MPP activated. Subjects experienced either an improvement, worsening, or no change in NYHA classification.
  The NYHA provides a simple way of classifying the extent of heart failure:
  NYHA I: No limitation of physical activity. Ordinary physical activity does not cause fatigue, palpitation, dyspnea.
  NYHA II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  NYHA III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  NYHA IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest.
Time Frame: 6 months
Population: Subjects implanted with a CRT-D device and a Quartet quadripolar LV lead, programmed with the MPP feature activated and who had a NYHA classification evaluation at baseline and 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | MPP ON
Number analyzed (Participants) | 82
Participants
  Improvement in NYHA classification | 26
  Worsening in NYHA classification | 2
  NYHA classification unchanged | 54

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Total Enrolled: All subjects enrolled in the study are included in the outcome measure.
Arm/Group | Total Enrolled
All-Cause Mortality (participants affected / at risk) | 2/105
Serious Adverse Events (participants affected / at risk) | 16/105
Other Adverse Events (participants affected / at risk) | 11/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Enrolled (N=105)
Atrial Arrhytmia (Cardiac disorders) | 2 (3)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Exacerbation of Heart Failure (Cardiac disorders) | 1 (1)
Trauma (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Inappropriate shock (Cardiac disorders) | 1 (1)
Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Lead dislodgment (Cardiac disorders) | 4 (6)
Pneumothorax/Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subclavian Vein Thrombus (Cardiac disorders) | 1 (1)
Twiddler´s Syndrome (Cardiac disorders) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Enrolled (N=105)
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma/Seratoma (Skin and subcutaneous tissue disorders) | 1 (1)
Inappropiate shock (Cardiac disorders) | 1 (1)
Intermittent pacing (Cardiac disorders) | 1 (1)
Lead dislodgement (Cardiac disorders) | 4 (4)
Oversensing (Cardiac disorders) | 1 (1)
Pectoral/Diaphragmatic/Phrenic Nerve Stimulation (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT02476201/Prot_SAP_000.pdf